CLINICAL TRIAL: NCT04873089
Title: RV3278AET0943 Cosmetic Product Efficacy Applied for 8 Weeks in Adults Having Oily and Acne Prone Skin: Comparative Study Versus Not Treated Group
Brief Title: Efficacy Study of Cosmetic Product RV3278AET0943 Versus Non-treated Group in Adults With Oily and Acne Prone Skin
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RV3278A2018243
Record Dates: First submitted 2021-04-21; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Acne
Keywords: Lipids; Biometrological; Microcomedomes; Sebum; Fatty acids; Phytotherapy
MeSH Terms: conditions — Acne Vulgaris | interventions — Cosmetics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Sebum and comedones constituents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RV3278A arm: RV3278A study product is applied twice a day (morning and evening) on the face during the whole study.
  Interventions: Other: Cosmetic product
- Control Group: Subjects included in the control group did not receive the test product or other associated product

INTERVENTIONS:
Other: Cosmetic product — It is a comparative study with two parallel groups of subjects:
  * Tested group: twice daily application of the cream RV3278A cosmetic product on the whole face
  * Comparative group: no application of study product or reference product
  Groups: RV3278A arm

SUMMARY:
The aim of this study is to evaluate, at different times, the RV3278A - ET0943 cosmetic product efficacy after 8 weeks of application on the face (twice-daily application). At T1 (Baseline), T2 (4 weeks) and T3 (8 weeks), the following assessments are performed:

* The reduction of the pilosebaceous follicular ostium size in vivo (pores) on the forehead
* The clinical evaluation (count of non inflammatory and inflammatory acne lesions, IGA score) of the face
* The reduction in visible follicles
* The standardized numerical photographs of face and ¾ right and left profile in normal, parallel polarized, cross polarized and UV light
* The analysis of the skin lipids of the forehead
* The qualitative and quantitative analysis of the sebum and comedones constituents (nose wings)

This is a comparative, open-labelled study, on subjects with oily and acne prone skins on the face.

Each group includes 18 subjects.

DETAILED DESCRIPTION:
This study is monocentric, comparative versus non-treated group, open-labelled, exploratory, conducted in adults having oily and acne prone skin.

The study includes 4 visits for each group, including subjects' selection:

* V0: Subjects' selection
* V1: Baseline inclusion
* V2: 4 weeks, follow-up visit
* V3: 8 weeks, study end

The maximal study duration is 61 days. The front, temporal areas and nose wings are defined as the study interest areas for superficial samples.

The evaluation is at 3 times: T1 baseline, T2 at 4 weeks and T3 at 8 weeks of application of RV3278A formula ET0943 with comparison of each time versus baseline.

There are twice-daily applications (morning and evening) of the test product on the face.

ELIGIBILITY:
Inclusion Criteria:

1. Criteria related to the population:

   * Male or Female aged between 18 and 35 years included
   * Subject with phototype I to IV included
   * Subject having signed his/her written informed consent for his/her participation in the study
   * Subject who is currently not participating in another clinical study
   * Subject affiliated to a social security system or health insurance, or is a beneficiary
   * For woman of childbearing potential: use of an effective method of contraception and using it during the whole duration of the study
2. Criteria related to diseases and general health:

   * Subject with oily, blemished skin and dilated pores on the face including open and closed comedones of the retention type (on the forehead, temporal areas and nose wings) and some inflammatory lesions:

     * Retention aspect: microcomedones and open comedones count on the forehead (> 10)
     * Inflammatory aspect: lesions ≤ 10 count on the whole face

Exclusion Criteria:

1. Criteria related to the population:

   * For woman of childbearing potential: subject pregnant or breastfeeding or planning to be pregnant during the study
   * Subject having already known allergy to latex
   * Subject having already known allergy to the test product or associated product components
   * Subject having scar(s) or other skin characteristic on the study areas (forehead, temporal areas and nose wings) and which, size is not compatible with the study realization
   * Subject who, has planned to apply exfoliating, keratolytic and/or self-tanning products on the face within 2 weeks prior to inclusion.
   * Subject who, has planned to be exposed to the natural or artificial UV during the study
   * Subject who is not likely to be compliant with study-related requirements
   * Subject deprived of freedom by administrative or legal decision or under guardianship
2. Criteria related to diseases and general health:

   - Inflammatory or immunological dermatosis (atopic dermatitis, psoriasis, severe inflammatory acne, cutaneous seborrhoeic dermatitis, vitiligo of the face..) of the face, or other dermatological face illness in progress at the time of inclusion on the sample areas (pigmentation of the sample areas by melasma, solar erythema or artificial post UV...)
3. Criteria related to treatments

   * Facial treatments :

     * Any topical anti-acne antibiotics (topical Erythromycin or topical Dalacin) applied during more than 5 consecutive days within 4 weeks before the inclusion
     * Any topical treatment (dermo corticoids, retinoids, antibiotics, antifungals…) ongoing or applied within 4 weeks before the inclusion
   * Oral intake of antibiotic, zinc gluconate or hormonal anti-acne treatments, ongoing or taken during more than 5 consecutive days within the month before the inclusion
   * Oral intake of isotretinoin within 6 months before the inclusion
   * Anti-inflammatory treatments (steroids or no steroids) according to the investigator's assessment
   * Hormonal contraception established or modified within 3 months before the inclusion
   * Application of skin care product containing exfoliating, keratolytic or self-tanning ingredients applied on the face within 15 days before the inclusion
   * Oral treatment (cardiovascular, endocrinal, rheumatological, urogenital, neuropsychiatric, immunosuppressant) established within 2 months before the inclusion not stabilized
   * Hygiene, skin care or make-up habits modified within less than one month before the inclusion

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects have been recruited from the panel of the centre. An investigator made a dermatological examination of the subjects before inscription in the panel. Data from this clinical examination, stored in the computer database with the consent of the subjects, can ensure the recruitment; computer software being questioned based on the eligibility criteria of the study.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Efficacy of the product on lesions count (Lucky method) | Change from baseline to 8 weeks later, for each group
  Inflammatory and lesions quantification on the whole face

SECONDARY OUTCOMES:
Efficacy of the product on lesions count (Lucky method) | Change from baseline to 4 weeks later, for each group
  Inflammatory and lesions quantification on the whole face
Forehead acne lesions count (target area) | Change from baseline to 4 weeks and 8 weeks later for each group, on the target area
Investigator Global Assessment (IGA) on 5-point scale | Change from 4 weeks to 8 weeks later, for each group, on the target area
  Clear = 0, Almost clear = 1, Mild = 2, Moderate = 3, Severe = 4
Sebum harvest and analysis | At baseline and after one month of tested product treatment
  Quantification of free fatty acid (FFA) / triglyceride (TG) ratio by infrared spectroscopy: Forehead sebum was collected on absorbent paper then the lipid composition was analysed by infrared spectroscopy to determine the free fatty acids to triglycerides ratio
Comedones lipid harvest and analysis | At baseline and after one month of tested product treatment
  Quantification of free fatty acid / triglyceride ratio by GC/MS: Samples were collected with patch on nose wings. Comedones were collected and lipids extracted according to the Bligh & Dyer (Bligh and Dyer, 1959). The biochemical exploration was performed by the screening of neutral lipids on GC/MS
Skin lipids | Change from baseline to 4 weeks and 8 weeks later, for each group, on the target area
  Measure by FTIR spectroscopy (in vivo non invasive infrared analysis)
Pilosebaceous follicular ostium size in vivo | Change from baseline to 4 weeks and 8 weeks later, for each group, on the target area
  Measure by confocal microscope
Dilated pores on 5-point scale | Change from baseline to 4 weeks and 8 weeks later, for each group, on the target area
  Absent = 0, Very mild = 1, Mild = 2, Moderate = 3, Severe = 4
Patient Global Assessment (PGA) on 6-points scale | Change from 4 weeks to 8 weeks later, for each group, on the target area
  Clear worsening = 0, slight worsening = 1, no change = 2, slight improvement = 3, clear improvement = 4, total improvement = 5
Self product agreement questionnaire | At week 8, for tested group
  9-question questionnaire with a majority of scales ranging from 0 to 10 where 0 was the worst satisfaction and 10 the best one
Visible follicles quantification by in vivo visualisation methods | Change from baseline to 4 weeks and 8 weeks later, for each group, on the target area
  Count by multispectral imaging

CONTACTS AND LOCATIONS:
Overall Officials: Thérèse NOCERA, MD dermatologist, Principal Investigator — SKIN RESEARCH CENTRE - Toulouse
Locations (1):
- Skin Research Centre, Toulouse, France

IPD SHARING:
Plan to Share IPD: No